CLINICAL TRIAL: NCT05632198
Title: UNCERTAINTY AS a BARRIER to SELF-CARE and QUALITY of LIFE in PATIENTS with HEART FAILURE with REDUCED EJECTION FRACTION
Brief Title: Uncertainty in HFrEF Patients
Status: Completed | Type: Observational
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Seyma Demir, Principal Investigator, Abant Izzet Baysal University
Other Study IDs: AIBU-HSF-SDEMIR-02
Record Dates: First submitted 2022-11-21; First posted 2022-11-30 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-07

CONDITIONS: Heart Failure with Reduced Ejection Fraction
Keywords: self care; quality of life; uncertainty
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Survey — Valid and reliable questionnaires covering perceived uncertainty, self-care behaviors and quality of life will be administered.

SUMMARY:
This study was planned as a descriptive and correlational type study to reveal the effect of perceived uncertainty by heart failure (HF) patients with reduced ejection fraction on quality of life and self-care behaviors. In this study, which aimed to reach 122 inpatients with HF, the dependent variables were quality of life and self-care behaviors, the independent variable will be perceived uncertainty. Data will be collected by Mishel Uncertainty in Illness Scale-Community Form (MUIS-C), Left Ventricular Disfunction Scale (LVD-36) and European Heart Failure Self-Care Behavior Scale (EHFSeBS). Data analysis will basically be done with Multivariate Analysis of Variance (MANOVA).

DETAILED DESCRIPTION:
This study aims to reveal the effect of perceived uncertainty on quality of life and self-care behaviors in HF patients with reduced ejection fraction. This descriptive and correlational study will include 122 HF patients hospitalized in the cardiology department of a university hospital in northern Turkey. The sample size was calculated according to parameters based on the power of 90%, 95% confidence interval, error level of 0.05, effect size of 0.59. Data will be collected by Mishel Uncertainty in Illness Scale-Community Form (MUIS-C), Left Ventricular Disfunction Scale (LVD-36) and European Heart Failure Self-Care Behavior Scale (EHFSeBS). Data analysis will basically be done with Multivariate Analysis of Variance (MANOVA).

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older,
* Having been diagnosed with heart failure by a physician for more than 6 months,
* Left ventricular ejection fraction <40% as measured by echocardiography,
* Volunteering in participating in the study

Exclusion Criteria:

* Being under antidepressant treatment,
* Presence of a pre-existing psychiatric illness or cognitive impairment,
* Diagnosed with cancer and being under treatment related to cancer,
* Presence of chronic obstructive pulmonary disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population identifies heart failure patients with reduced ejection fraction (< %40) as evidenced by an echocardiogram.
Sampling Method: Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2024-06-11 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
Uncertainty (questionnaire) | Baseline
  Mishel Uncertainty in Illness Scale-Community Form (MUIS-C) will be used to measure perceived uncertainty. The 20-item Turkish version of the scale has three sub-dimensions: Perception of the current situation (Cronbach's alpha = 0.86), perception of understanding (Cronbach's alpha = 0.78), ambiguity (Cronbach's alpha = 0.79). The total score is obtained by adding the scores given to each item of the five-point Likert scale. Thus, the score that can be obtained from the scale varies between 20 and 100, with an average of 60. An increase in the score obtained from the scale is interpreted as an increase in perceived uncertainty. Cronbach's alpha coefficients calculated in different HF populations using the scale ranged from 0.79 to 0.92, including the Turkish version.
Quality of life (questionnaire) | Baseline
  Left Ventricule Disfunction Scale (LVD-36) will be used to measure quality of life. The 36-item Turkish version of the scale consists of 36 items and the questions are presented to the patients with two options as true or false. The correct answers given are added together and the total number of correct answers found is expressed as a percentage. Scores between 0 and 100 are taken from the scale, and as the score increases, the quality of life decreases.Cronbach's alpha coefficient of the Turkish version of the scale was calculated as 0.87.
Self-care behavior (questionnaire) | Baseline
  European Heart Failure Self-Care Behavior Scale (EHFSeBS) will be used to measure self-care behavior. The scale is a 5-point Likert scale consisting of 12 questions that measures the definition of symptoms such as edema, respiratory distress, and fatigue related to HF, regular use of medications for these symptoms, fluid and salt restriction, communication with health personnel, and self-care assessment actions such as weight monitoring. The total score that can be obtained from the scale varies between 12-60. A high total score indicates low self-care, and a low score indicates high self-care. Cronbach's alpha coefficient of the Turkish version of the scale was calculated as 0.69.

CONTACTS AND LOCATIONS:
Overall Officials: Şeyma Demir Erbaş, PhD, Principal Investigator — Bolu Abant Izzet Baysal University, Faculty of Health Sciences
Locations (1):
- Bolu Abant Izzet Baysal University, Bolu, Bolu, Turkey (Türkiye)